CLINICAL TRIAL: NCT01863329
Title: Comparison of Optic Nerve Sheath Diameter on Retrobulbar Ultrasound Before and After Drainage of Cerebrospinal Fluid in Patient With Hydrocephalus
Status: Terminated | Type: Observational
Why Stopped: The investigator resigned on February 28, 2014.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0006
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2014-12

CONDITIONS: Hydrocephalus
Keywords: Optic nerve sheath diameter; Hydrocephalus; Intracranial hypertension
MeSH Terms: conditions — Hydrocephalus; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- both optic nerve sheath diameter: both optic nerve sheath diameter (the posterior 3mm of the papilla), 5 individual measurement
  Interventions: Procedure: retrobulbar ultrasound

INTERVENTIONS:
Procedure: retrobulbar ultrasound — both optic nerve sheath diameter (the posterior 3mm of the papilla), 5 individual measurement

SUMMARY:
Studies in patients with intracranial hypertension have shown a good relationship between optic nerve sheath diameter measured by retrobulbar ultrasound and invasively measured intracranial pressure. The aim of this study was to evaluate changes in optic nerve sheath diameter before and after drainage of cerebrospinal fluid in patients with hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ-Ⅱ
2. aged between 20 and 70 year
3. hydrocephalus
4. general anesthesia for undergoing drainage of cerebrospinal fluid

Exclusion Criteria:

1. an anatomical or functional abnormality in optic nerve

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
both optic nerve sheath diameter (the posterior 3mm of the papilla) | from induction of general anesthesia to average 15 min after recovery of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea